CLINICAL TRIAL: NCT01870869
Title: NATRELLE® 410 X-Style and L-Style Breast Implants Continued Access Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There was no indication that long-term follow-up would differ between any of the studies that have evaluated devices within the 410 Style Matrix.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 410CAXL-001
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Breast Augmentation; Breast Reconstruction; Breast Implant Revision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (4):
- Augmentation (Experimental): Women who had breast augmentation with NATRELLE® 410 implants.
  Interventions: Device: Anatomically shaped, silicone-filled breast implants with low height/projection or extra-full projection
- Reconstruction (Experimental): Women who had breast reconstruction with NATRELLE® 410 implants.
  Interventions: Device: Anatomically shaped, silicone-filled breast implants with low height/projection or extra-full projection
- Revision-Augmentation (Experimental): Women who had revision of previous breast augmentation with NATRELLE® 410 implants.
  Interventions: Device: Anatomically shaped, silicone-filled breast implants with low height/projection or extra-full projection
- Revision-Reconstruction (Experimental): Women who had revision of previous breast reconstruction with NATRELLE® 410 implants.
  Interventions: Device: Anatomically shaped, silicone-filled breast implants with low height/projection or extra-full projection

INTERVENTIONS:
Device: Anatomically shaped, silicone-filled breast implants with low height/projection or extra-full projection — Surgical implant
  Other Names: NATRELLE® 410 Highly Cohesive Anatomically Shaped Silicone-Filled Breast Implants (Styles FX, MX, LX, FL, ML, LL, LM, and LF)

SUMMARY:
This study is a prospective, multicenter, nonrandomized study to provide access to and evaluate the safety and effectiveness of NATRELLE® 410 Highly Cohesive Anatomically Shaped Silicone-Filled X-Style and L-Style Breast Implants for breast augmentation, reconstruction, or revision.

ELIGIBILITY:
Inclusion Criteria:

For entry in this study, participants must have either been enrolled in the 410 CA Clinical Study or 410 CARE Clinical Study under the inclusion criteria below and received NATRELLE® 410 Highly Cohesive Anatomically Shaped Silicone-Filled X- or L-Style Breast Implants in 1 or both breasts; or be planning to be implanted with NATRELLE® 410 Highly Cohesive Anatomically Shaped Silicone-Filled X- or L-Style Breast Implants in 1 or both breasts and meet the inclusion criteria listed below:

* Female, age 18 or older (age 22 or older for breast augmentation participants who are implanted under Protocol 410CAXL-001)
* Present with 1 or more of the following conditions:

  * Primary breast augmentation (i.e., no previous breast implant surgery) indicated for participant dissatisfaction with size or shape of breast (e.g., mammary hypoplasia), asymmetry, ptosis, or aplasia
  * Primary breast reconstruction (i.e., no previous breast implant surgery other than implantation of tissue expanders or contralateral augmentation for asymmetry) indicated, in the affected breast, for mastectomy for cancer, prophylactic mastectomy, or breast trauma, (resulting in mastectomy) and for the unaffected breast, contralateral asymmetry (may be performed on the date of the mastectomy or the date when permanent implants are placed in the reconstructed breast)
  * Breast implant revision surgery (i.e., removal and replacement of breast implants) indicated for previous augmentation or reconstruction with silicone-filled or saline-filled breast implants
* Has adequate tissue available to cover implants

Exclusion Criteria:

For entry in this study, participants must have either been enrolled in the 410 CA Clinical Study or 410 CARE Clinical Study and did not meet the exclusion criteria listed below or plan to undergo implantation with NATRELLE® 410 Highly Cohesive Anatomically Shaped Silicone-Filled X- or L-Style Breast Implants in 1 or both breasts and does not meet the exclusion criteria listed below:

* Has an advanced fibrocystic disease considered to be premalignant without accompanying subcutaneous mastectomy
* Has an existing carcinoma of the breast, without mastectomy
* Has an abscess or infection in the body at the time of enrollment
* Is pregnant or nursing
* Has any disease, including uncontrolled diabetes (e.g., hemoglobin A1c (HbA1c) > 8%), that is clinically known to impact wound healing ability
* Shows tissue characteristics that are clinically incompatible with mammaplasty, such as tissue damage resulting from radiation, inadequate tissue, compromised vascularity, or ulceration
* Has or is under treatment for any condition that may constitute an unwarranted surgical risk (e.g., unstable cardiac or pulmonary problems)
* Shows psychological characteristics that may be incompatible with the surgical procedure and the prosthesis, such as inappropriate attitude or motivation (e.g., body dysmorphic disorder)
* Is not willing to undergo further surgery for revision, if medically required

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1951 (Actual)
Dates: Start 2013-05-29 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Schumacher, Study Chair — Allergan
Locations (57):
- United States (57):
  - Anthony Griffin, Beverly Hills, California
  - Laurence Berkowitz, Campbell, California
  - Mary Powers, Long Beach, California
  - Roy Hong, Palo Alto, California
  - Eric Bachelor, Pleasanton, California
  - Douglas Reavie, San Diego, California
  - Steven Teitelbaum, Santa Monica, California
  - Tad Heinz, Colorado Springs, Colorado
  - Gary Snider, Denver, Colorado
  - Terrence Murphy, Englewood, Colorado
  - Orlando De Lucia, Farmington, Connecticut
  - Lewis Berger, Tampa, Florida
  - Gerard Mosiello, Tampa, Florida
  - James Namnoum, Atlanta, Georgia
  - Peter Johnson, Des Plaines, Illinois
  - Stephen Madry, Elk Grove Village, Illinois
  - Janet Turkle, Carmel, Indiana
  - Bruce Van Natta, Indianapolis, Indiana
  - Christine Kelley-Patteson, Indianapolis, Indiana
  - Brad Storm, Olathe, Kansas
  - Julene Samuels, Louisville, Kentucky
  - Timothy Mickel, Monroe, Louisiana
  - Paul Davis, Shreveport, Louisiana
  - Bradley Bengtson, Grand Rapids, Michigan
  - John Renucci, Grand Rapids, Michigan
  - Steven Morris, Midland, Michigan
  - Charles Nathan, Chesterfield, Missouri
  - Herluf Lund Jr., Chesterfield, Missouri
  - Patricia McGuire, Creve Coeur, Missouri
  - Schuyler Meltis, Hannibal, Missouri
  - Perry Johnson, Omaha, Nebraska
  - Peter Hyans, Berkeley Heights, New Jersey
  - Isaac Starker, Florham Park, New Jersey
  - Peter Hetzler, Little Silver, New Jersey
  - Marc Alan Drimmer, Princeton, New Jersey
  - Caroline Glicksman, Sea Girt, New Jersey
  - Lloyd Gayle, New York, New York
  - John Sherman, New York, New York
  - Tracy Pfeifer, New York, New York
  - Robert Jacobs, Port Jefferson Station, New York
  - John Decorato, Staten Island, New York
  - Raymond Isakov, Cleveland, Ohio
  - Craig Colville, Toledo, Ohio
  - Frank Barone, Toledo, Ohio
  - Derek Shadid, Oklahoma City, Oklahoma
  - Robert Hein, Oklahoma City, Oklahoma
  - Mark Jewell, Eugene, Oregon
  - John Lettieri, Spartanburg, South Carolina
  - Kristina D. O'Shaughnessy, Nashville, Tennessee
  - Patrick Maxwell, Nashville, Tennessee
  - William Carpenter, Dallas, Texas
  - Jeffrey Friedman, Houston, Texas
  - Natan Yaker, Plano, Texas
  - William Adams, University Park, Texas
  - Gloria Duda, McLean, Virginia
  - Gavin Dry, Bellevue, Washington
  - Allen Gabriel, Vancouver, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Started | 288 | 206 | 1222 | 235
Completed | 260 | 192 | 1092 | 205
Not Completed | 28 | 14 | 130 | 30
Not completed — Implanted with nonstudy device | 1 | 3 | 14 | 4
Not completed — Death | 0 | 0 | 7 | 1
Not completed — Subject choice | 6 | 2 | 22 | 8
Not completed — Lost to Follow-up | 10 | 2 | 25 | 3
Not completed — Reason not Specified | 1 | 2 | 20 | 4
Not completed — Not evaluable | 10 | 5 | 42 | 10

BASELINE CHARACTERISTICS:
Population: Evaluable population was defined as all participants enrolled under this study protocol who received a NATRELLE® 410 X- or L-style device.
Groups:
- Total: Total of all reporting groups
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction | Total
Number analyzed (Participants) | 278 | 201 | 1180 | 225 | 1884
Age, Continuous [Mean (Full Range); unit: years] — Population: Number analyzed is the number of participants with available age data.
  years
    number analyzed (Participants) | 277 | 201 | 1176 | 223 | 1877
    (all) | 34.5 [18.0 to 63.0] | 47.3 [20.0 to 79.0] | 50.3 [21.0 to 79.0] | 54.4 [31.0 to 80.0] | 48.1 [18.0 to 80.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 278 | 201 | 1180 | 225 | 1884
  Male | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants According to Investigator Satisfaction With Implants
Description: The investigator rated their satisfaction with the participant's breast implant for each breast on a 5-point scale (1=Definitely dissatisfied, 2=Somewhat dissatisfied, 3=Neither satisfied or dissatisfied, 4=Somewhat satisfied, 5=Definitely satisfied). If there was a different response for the left and right breasts the worst response was used. The percentage of participants where the investigator responded: "Definitely satisfied" or "Somewhat satisfied" is reported.
Time Frame: 5 years (followup after implantation that occurred between 06 May 2008 and 08 January 2015)
Population: Participants from the Evaluable population, all participants enrolled under this study protocol who received a NATRELLE® 410 X- or L-style device, with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 77 | 34 | 247 | 52
percentage of participants
  Definitely satisfied | 94.8 | 85.3 | 74.1 | 73.1
  Somewhat satisfied | 3.9 | 8.8 | 21.5 | 23.1

2. Primary Outcome: Percentage of Participants According to Participant Satisfaction With Implants
Description: The participant rated their satisfaction with the breast implant for each breast on a 5-point scale (1=Definitely dissatisfied, 2=Somewhat dissatisfied, 3=Neither satisfied or dissatisfied, 4=Somewhat satisfied, 5=Definitely satisfied). If there was a different response for the left and right breasts the worst response was used. The percentage of participants who responded: "Definitely satisfied" or "Somewhat satisfied" is reported.
Time Frame: 5 years (followup after implantation that occurred between 06 May 2008 and 08 January 2015)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 77 | 34 | 247 | 52
percentage of participants
  Definitely satisfied | 88.3 | 76.5 | 68.0 | 65.4
  Somewhat satisfied | 5.2 | 17.6 | 24.7 | 25.0

3. Secondary Outcome: Percentage of Participants With Local Complications
Description: Kaplan-Meier risk rates (estimation of the percentage of participants) of developing local complications is presented. Local complications collected in the study were: Asymmetry, Breast pain, Capsular contracture, Delayed wound healing, Fluid accumulation/seroma, Hematoma, Hypertrophic scarring/other abnormal scarring, Implant extrusion, Implant malposition, Implant palpability/visibility, Implant rupture, Infection, Redness, Skin rash, Swelling, Tissue/skin necrosis, Upper pole fullness, Wrinkling/rippling and Other complications .
Time Frame: 5 years (followup after implantation that occurred between 06 May 2008 and 08 January 2015)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 278 | 201 | 1180 | 225
percentage of participants
  Any complication | 6.62 [3.78 to 11.45] | 9.09 [5.65 to 14.46] | 14.50 [11.78 to 17.78] | 10.19 [6.81 to 15.11]
  Asymmetry | 1.11 [0.26 to 4.73] | 1.99 [0.75 to 5.21] | 2.34 [1.59 to 3.44] | 2.67 [1.21 to 5.84]
  Breast pain | 1.93 [0.51 to 7.15] | 1.08 [0.15 to 7.39] | 0.51 [0.23 to 1.13] | 1.07 [0.26 to 4.30]
  Capsular contracture | 1.85 [0.68 to 4.98] | 7.90 [3.57 to 17.01] | 20.14 [8.90 to 41.85] | 27.03 [9.04 to 64.93]
  Delayed wound healing | 0.00 [0.00 to 0.00] | 0.50 [0.07 to 3.48] | 0.34 [0.13 to 0.90] | 1.78 [0.67 to 4.67]
  Fluid accumulation/seroma | 0.37 [0.05 to 2.57] | 0.50 [0.07 to 3.48] | 0.57 [0.26 to 1.28] | 1.78 [0.67 to 4.67]
  Hematoma | 0.00 [0.00 to 0.43] | 0.00 [0.00 to 0.00] | 0.43 [0.18 to 1.04] | 0.44 [0.06 to 3.11]
  Hypertrophic scarring/other abnormal scarring | 0.72 [0.18 to 2.85] | 1.29 [0.32 to 5.12] | 0.75 [0.24 to 2.30] | 0.44 [0.06 to 3.11]
  Implant extrusion | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.98 [0.40 to 2.38] | 0.60 [0.08 to 4.17]
  Implant malposition | 2.21 [0.80 to 6.07] | 1.00 [0.25 to 3.92] | 1.22 [0.52 to 2.84] | 1.33 [0.43 to 4.08]
  Implant palpability/visibility | 0.48 [0.07 to 3.33] | 0.00 [0.00 to 0.00] | 0.25 [0.08 to 0.79] | 0.44 [0.06 to 3.11]
  Implant rupture | 2.14 [0.67 to 6.75] | 6.15 [1.77 to 20.22] | 2.03 [0.91 to 4.50] | 3.84 [1.39 to 10.38]
  Infection | 0.36 [0.05 to 2.53] | 1.49 [0.48 to 4.56] | 1.21 [0.72 to 2.04] | 3.18 [1.53 to 6.56]
  Redness | 0.00 [0.00 to 0.00] | 0.50 [0.07 to 3.48] | 0.83 [0.29 to 2.38] | 3.31 [1.01 to 10.59]
  Skin rash | 0.36 [0.05 to 2.53] | 0.00 [0.00 to 0.00] | 0.08 [0.01 to 0.60] | 0.00 [0.00 to 0.00]
  Swelling | 0.72 [0.18 to 2.85] | 0.00 [0.00 to 0.00] | 0.17 [0.04 to 0.68] | 0.44 [0.06 to 3.11]
  Tissue/skin necrosis | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.17 [0.04 to 0.68] | 0.50 [0.07 to 3.51]
  Upper pole fullness | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.44 [0.06 to 3.11]
  Wrinkling/rippling | 0.00 [0.00 to 0.00] | 0.50 [0.07 to 3.48] | 1.61 [0.78 to 3.33] | 0.00 [0.00 to 0.00]
  Other complications | 1.46 [0.45 to 4.70] | 2.99 [1.35 to 6.52] | 4.37 [2.94 to 6.46] | 1.43 [0.46 to 4.38]

4. Secondary Outcome: Percentage of Participants With Reoperations
Description: Kaplan-Meier risk rates (estimation of the percentage of participants) of reoperation is reported.
Time Frame: 5 years (followup after implantation that occurred between 06 May 2008 and 08 January 2015)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 278 | 201 | 1180 | 225
percentage of participants | 13.02 [8.42 to 19.84] | 25.08 [16.99 to 36.09] | 39.70 [35.35 to 44.38] | 35.75 [27.42 to 45.72]

5. Secondary Outcome: Percentage of Participants With Implant Removal With or Without Replacement
Description: Kaplan-Meier risk rates (estimation of the percentage of participants) of implant removal with or without replacement is reported.
Time Frame: 5 years (followup after implantation that occurred between 06 May 2008 and 08 January 2015)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Number analyzed (Participants) | 278 | 201 | 1180 | 225
percentage of participants | 7.17 [3.80 to 13.31] | 19.09 [11.12 to 31.66] | 19.54 [15.79 to 24.03] | 20.59 [13.59 to 30.50]

ADVERSE EVENTS:
Time Frame: 5 years (followup after implantation that occurred between 06 May 2008 and 08 January 2015)
Description: Adverse events were not collected in this study. Deaths are reported as Serious Adverse Events. Specific local complications were collected and are reported in the Outcome Measure section. Evaluable population.
Arm/Group | Augmentation | Revision-Augmentation | Reconstruction | Revision-Reconstruction
Serious Adverse Events (participants affected / at risk) | 0/278 | 0/201 | 7/1180 | 1/225
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Augmentation (N=278) | Revision-Augmentation (N=201) | Reconstruction (N=1180) | Revision-Reconstruction (N=225)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Metastatic carcinoma to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Recurrence of breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Liver cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastatic breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.